CLINICAL TRIAL: NCT04492475
Title: A Multicenter, Adaptive, Randomized Blinded Controlled Trial of the Safety and Efficacy of Investigational Therapeutics for the Treatment of COVID-19 in Hospitalized Adults (ACTT-3)
Brief Title: Adaptive COVID-19 Treatment Trial 3 (ACTT-3)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-0006 ACTT-3
Record Dates: First submitted 2020-07-28; First posted 2020-07-30 (Actual); Results first posted 2021-11-22 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2020-11

CONDITIONS: COVID-19
Keywords: Adaptive; COVID-19; Efficacy; Multicenter; novel coronavirus; Safety
MeSH Terms: conditions — COVID-19 | interventions — Interferon beta-1a; remdesivir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Remdesivir plus Interferon Beta-1a (Experimental): 200 mg of Remdesivir administered intravenously on Day 1, followed by a 100 mg once-daily maintenance dose of Remdesivir while hospitalized for up to a 10-day total course and 44 mcg of interferon beta-1a administered by a 0.5 mL subcutaneous injection on Days 1, 3, 5, and 7 while hospitalized for a total of 4 doses.
  Interventions: Drug: Interferon beta-1a; Drug: Remdesivir
- Remdesivir plus Placebo (Placebo Comparator): 200 mg of Remdesivir administered intravenously on Day 1, followed by a 100 mg once-daily maintenance dose of Remdesivir while hospitalized for up to a 10-day total course and a 0.5 mL placebo injection administered subcutaneously on Days 1, 3, 5, and 7 while hospitalized for a total of 4 doses.
  Interventions: Other: Placebo; Drug: Remdesivir

INTERVENTIONS:
Drug: Interferon beta-1a — Rebif (R) is a purified 166 amino acid human interferon beta glycoprotein with an amino acid sequence identical to natural fibroblast derived human interferon beta. Each 0.5 mL prefilled syringe contains 44 mcg of interferon beta-1a, 4 mg human albumin, USP; 27.3 mg mannitol, USP; 0.4 mg sodium acetate; and water for injection, USP.
  Arms: Remdesivir plus Interferon Beta-1a
Other: Placebo — The interferon beta-1a placebo contains either 0.5 mL 0.9% normal saline or 0.5 mL sterile water for injection.
  Arms: Remdesivir plus Placebo
Drug: Remdesivir — Drug Remdesivir is a single diastereomer monophosphoramidate prodrug designed for the intracellular delivery of a modified adenine nucleoside analog GS-441524. In addition to the active ingredient, the lyophilized formulation of Remdesivir contains the following inactive ingredients: water for injection, sulfobutylether beta-cyclodextrin sodium (SBECD), and hydrochloric acid and/or sodium hydroxide.

SUMMARY:
ACTT-3 will evaluate the combination of interferon beta-1a and remdesivir compared to remdesivir alone. Subjects will be assessed daily while hospitalized. If the subjects are discharged from the hospital, they will have a study visit at Days 15, 22, and 29. For discharged subjects, it is preferred that the Day 15 and 29 visits are in person to obtain safety laboratory tests and oropharyngeal (OP) swab and blood (serum only) samples for secondary research as well as clinical outcome data. However, infection control or other restrictions may limit the ability of the subject to return to the clinic. In this case, these visits may be conducted by phone, and only clinical data will be obtained. The Day 22 visit does not have laboratory tests or collection of samples and is conducted by phone. The primary outcome is time to recovery by Day 29.

DETAILED DESCRIPTION:
This study is an adaptive randomized double-blind placebo-controlled trial to evaluate the safety and efficacy of novel therapeutic agents in hospitalized adults diagnosed with COVID-19. The study is a multicenter trial that will be conducted in up to approximately 100 sites globally. The study will compare different investigational therapeutic agents to a control arm. New arms can be introduced according to scientific and public health needs. There will be interim monitoring to allow early stopping for futility, efficacy, or safety. If one therapy proves to be efficacious, then this treatment may become the control arm for comparison(s) with new experimental treatment(s). Any such change would be accompanied by an updated sample size. This adaptive platform is used to rapidly evaluate different therapeutics in a population of those hospitalized with moderate to severe COVID-19. The platform will provide a common framework sharing a similar population, design, endpoints, and safety oversight. New stages with new therapeutics can be introduced. One independent Data and Safety Monitoring Board (DSMB) will actively monitor interim data in all stages to make recommendations about early study closure or changes to study arms.

ACTT-3 will evaluate the combination of interferon beta-1a and remdesivir compared to remdesivir alone. Subjects will be assessed daily while hospitalized. If the subjects are discharged from the hospital, they will have a study visit at Days 15, 22, and 29. For discharged subjects, it is preferred that the Day 15 and 29 visits are in person to obtain safety laboratory tests and oropharyngeal (OP) swab and blood (serum only) samples for secondary research as well as clinical outcome data. However, infection control or other restrictions may limit the ability of the subject to return to the clinic. In this case, these visits may be conducted by phone, and only clinical data will be obtained. The Day 22 visit does not have laboratory tests or collection of samples and is conducted by phone.

All subjects will undergo a series of efficacy, safety, and laboratory assessments. Safety laboratory tests and blood (serum and plasma) research samples and oropharyngeal (OP) swabs will be obtained on Days 1 (prior to infusion) and Days 3, 5, 8, and 11 (while hospitalized). OP swabs and blood (serum only) plus safety laboratory tests will be collected on Day 15 and 29 (if the subject attends an in-person visit or are still hospitalized).

The primary outcome is time to recovery by Day 29 for patients with baseline ordinal score 4, 5 and 6. A key secondary outcome evaluates treatment-related improvements in the 8-point ordinal scale at Day 15. Each stage may prioritize different secondary endpoints for the purpose of multiple comparison analyses.

Contacts:

20-0006 Central Contact

Telephone: 1 (301) 7617948

Email: DMIDClinicalTrials@niaid.nih.gov

ELIGIBILITY:
Inclusion Criteria:

1. Admitted to a hospital with symptoms suggestive of COVID-19.
2. Subject (or legally authorized representative) provides informed consent prior to initiation of any study procedures.
3. Subject (or legally authorized representative) understands and agrees to comply with planned study procedures.
4. Male or non-pregnant female adult > / = 18 years of age at time of enrollment.
5. Has laboratory-confirmed SARS-CoV-2 infection as determined by polymerase chain reaction (PCR) or other commercial or public health assay in any respiratory specimen or saliva, as documented by either of the following:

   * PCR or other assay positive in sample collected < 72 hours prior to randomization; OR
   * PCR or other assay positive in sample collected >/= 72 hours but < 7 days prior to randomization AND progressive disease suggestive of ongoing SARS-CoV-2 infection.

   Note: if written documentation of the positive test result is not available at enrollment (e.g., report from other institution), the subject may be enrolled but the PCR should be repeated at the time of enrollment.
6. Illness of any duration, and at least one of the following:

   * Radiographic infiltrates by imaging (chest x-ray, CT scan, etc.), OR
   * SpO2 < / = 94% on room air, OR
   * Requiring supplemental oxygen.
7. Women of childbearing potential must agree to either abstinence or use at least one primary form of contraception not including hormonal contraception from the time of screening through Day 29.
8. Agrees to not participate in another clinical trial (both pharmacologic and other types of interventions) for the treatment of COVID-19 through Day 29.

Exclusion Criteria:

1. Anticipated discharge from the hospital or transfer to another hospital which is not a study site within 72 hours.
2. Subject meets criteria for ordinal scale category 6 or 7 at the time of screening.
3. Subject has a positive test for influenza virus during this current hospital admission.
4. Subjects with an estimated glomerular filtration rate (eGFR) < 30 mL/min are excluded unless in the opinion of the PI, the potential benefit of receiving remdesivir outweighs the potential risk of study participation.
5. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 times the upper limits of normal.
6. Total white cell blood cell count (WBC) <1500 cells/microliter.
7. Platelet count <50,000/microliter.
8. History of chronic liver disease (e.g., jaundice, ascites, hepatic encephalopathy, history of bleeding esophageal or gastric varices). No laboratory testing is needed.
9. Pregnancy or breast feeding (lactating women who agree to discard breast milk from Day 1 until three weeks after the last study product is given are not excluded).
10. Allergy to any study medication including history of hypersensitivity to natural or recombinant interferon beta or human albumin.
11. Patient has a chronic or acute medical condition or is taking a medication that cannot be discontinued at enrollment, that in the judgement of the PI, places them at unacceptable risk for a poor clinical outcome if they were to participate in the study.
12. Received three or more doses of remdesivir, including the loading dose, outside of the study for COVID-19.
13. Received convalescent plasma or intravenous immunoglobulin [IVIg] for the treatment of COVID-19.
14. Received any interferon product within two weeks of screening, either for the treatment of COVID-19 or for a chronic medical condition (e.g., multiple sclerosis, HCV infection).
15. Received any of the following in the two weeks prior to screening as treatment of COVID-19:

    * Small molecule tyrosine kinase inhibitors (e.g. baricitinib, imatinib, gefitinib, acalabrutinib, etc.);
    * Monoclonal antibodies targeting cytokines (e.g., TNF inhibitors, anti-interleukin-1 [IL-1], anti-IL-6 [tocilizumab or sarilumab], etc.);
    * Monoclonal antibodies targeting T-cells or B-cells as treatment for COVID-19.
16. Prior enrollment in ACTT-3.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 969 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2020-12-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (64):
- United States (55):
  - University of Alabama at Birmingham School of Medicine - Infectious Disease, Birmingham, Alabama
  - UCSF Fresno Center for Medical Education and Research - Clinical Research Center, Fresno, California
  - University of California San Diego Health - Jacobs Medical Center, La Jolla, California
  - University of California Los Angeles Medical Center - Westwood Clinic, Los Angeles, California
  - University of California Irvine Medical Center - Infectious Disease, Orange, California
  - VA Palo Alto Health Care System - Infectious Diseases, Palo Alto, California
  - Stanford University - Stanford Hospital and Clinics - Pediatrics - Infectious Diseases, Palo Alto, California
  - University of California Davis Medical Center - Internal Medicine - Infectious Disease, Sacramento, California
  - Naval Medical Center San Diego - Infectious Disease Clinic, San Diego, California
  - University of California San Francisco - Zuckerberg San Francisco General Hospital - Division of HIV, ID, and Global Medicine, San Francisco, California
  - Cedars Sinai Medical Center, West Hollywood, California
  - Eastern Colorado Health Care System, Aurora, Colorado
  - Denver Health Division of Hospital Medicine - Main Campus, Denver, Colorado
  - University of Florida Health - Shands Hospital - Division of Infectious Diseases and Global Medicine, Gainesville, Florida
  - University of Florida Health - Jacksonville - Department of Emergency Medicine, Jacksonville, Florida
  - University of Miami Miller School of Medicine - Infectious Diseases, Miami, Florida
  - Emory Vaccine Center - The Hope Clinic, Decatur, Georgia
  - Atlanta VA Medical Center - Infectious Diseases Clinic, Decatur, Georgia
  - Tripler Army Medical Center (TAMC), Honolulu, Hawaii
  - Northwestern Hospital - Infectious Disease, Chicago, Illinois
  - University of Illinois at Chicago Division of Infectious Diseases, Chicago, Illinois
  - University of Iowa Hospitals & Clinics - Department of Internal Medicine, Iowa City, Iowa
  - Ochsner Medical Center - Kenner - Department of Infectious Diseases, Kenner, Louisiana
  - Southeast Louisiana Veterans Health Care System - Section of Infectious Diseases, New Orleans, Louisiana
  - University of Maryland School of Medicine - Center for Vaccine Development - Baltimore, Baltimore, Maryland
  - Johns Hopkins Hospital - Medicine - Infectious Diseases, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - National Institutes of Health - Clinical Center, National Institute of Allergy and Infectious Diseases Laboratory Of Immunoregulation, Clinical Research Section, Bethesda, Maryland
  - Massachusetts General Hospital - Infectious Diseases, Boston, Massachusetts
  - University of Massachusetts Medical School - Infectious Diseases and Immunology, Worcester, Massachusetts
  - University of Minnesota Medical Center, Fairview - Infectious Diseases and International Medicine, Minneapolis, Minnesota
  - Saint Louis University - Center for Vaccine Development, St Louis, Missouri
  - University of Nebraska Medical Center - Infectious Diseases, Omaha, Nebraska
  - University of New Mexico Clinical and Translational Science Center, Albuquerque, New Mexico
  - New York University School of Medicine - Langone Medical Center - Microbiology - Parasitology, New York, New York
  - University of Rochester Medical Center - Vaccine Research Unit, Rochester, New York
  - Montefiore Medical Center - Infectious Diseases, The Bronx, New York
  - Duke Human Vaccine Institute - Duke Vaccine and Trials Unit, Durham, North Carolina
  - Womack Army Medical Center - Pulmonary and Respiratory Services, Fort Bragg, North Carolina
  - Kaiser Permanente Northwest - Center for Health Research, Portland, Oregon
  - Penn State Health Milton S. Hershey Medical Center - Division of Infectious Diseases, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania - Infectious Diseases, Philadelphia, Pennsylvania
  - Baylor Scott & White Health - Baylor University Medical Center - North Texas Infectious Disease Consultants, Dallas, Texas
  - University of Texas Southwestern Medical Center - Internal Medicine - Infectious Diseases, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch - Division of Infectious Disease, Galveston, Texas
  - Baylor College of Medicine - Molecular Virology and Microbiology, Houston, Texas
  - Methodist Hospital - Houston, Houston, Texas
  - University of Texas Health Science Center at San Antonio - Infectious Diseases, San Antonio, Texas
  - University of Utah - Infectious Diseases, Salt Lake City, Utah
  - University of Virginia - Acute Care Surgery, Charlottesville, Virginia
  - Naval Medical Center Portsmouth - Infectious Disease Division, Portsmouth, Virginia
  - EvergreenHealth Infectious Disease Service, Kirkland, Washington
  - Providence Sacred Heart Medical Center, Spokane, Washington
  - Madigan Army Medical Center - Infectious Disease Clinic, Tacoma, Washington
- National Center for Global Health and Medicine Hospital - Disease Control and Prevention Center, Tokyo, Japan
- Mexico (2):
  - Instituto Nacional de Enfermedades Respiratorias (INER) - Ismael Cosío Villegas, Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutrición Salvador Zubirán - Departamento de Infectologia, Mexico City
- Singapore (4):
  - National University Health System - Division of Infectious Diseases, Singapore
  - National Centre for Infectious Diseases (NCID), Singapore
  - Changi General Hospital - Clinical Trials and Research Unit (CTRU), Singapore
  - Ng Teng Fong General Hospital - Infectious Disease Service, Singapore
- South Korea (2):
  - Seoul National University Bundang Hospital - Division of Infectious Diseases, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul, Jongno-gu

REFERENCES:
- [Derived] Potter GE, Bonnett T, Rubenstein K, Lindholm DA, Rapaka RR, Doernberg SB, Lye DC, Mularski RA, Hynes NA, Kline S, Paules CI, Wolfe CR, Frank MG, Rouphael NG, Deye GA, Sweeney DA, Colombo RE, Davey RT Jr, Mehta AK, Whitaker JA, Castro JG, Amin AN, Colombo CJ, Levine CB, Jain MK, Maves RC, Marconi VC, Grossberg R, Hozayen S, Burgess TH, Atmar RL, Ganesan A, Gomez CA, Benson CA, Lopez de Castilla D, Ahuja N, George SL, Nayak SU, Cohen SH, Lalani T, Short WR, Erdmann N, Tomashek KM, Tebas P. Temporal Improvements in COVID-19 Outcomes for Hospitalized Adults: A Post Hoc Observational Study of Remdesivir Group Participants in the Adaptive COVID-19 Treatment Trial. Ann Intern Med. 2022 Dec;175(12):1716-1727. doi: 10.7326/M22-2116. Epub 2022 Nov 29. PMID 36442063
- [Derived] Kalil AC, Mehta AK, Patterson TF, Erdmann N, Gomez CA, Jain MK, Wolfe CR, Ruiz-Palacios GM, Kline S, Regalado Pineda J, Luetkemeyer AF, Harkins MS, Jackson PEH, Iovine NM, Tapson VF, Oh MD, Whitaker JA, Mularski RA, Paules CI, Ince D, Takasaki J, Sweeney DA, Sandkovsky U, Wyles DL, Hohmann E, Grimes KA, Grossberg R, Laguio-Vila M, Lambert AA, Lopez de Castilla D, Kim E, Larson L, Wan CR, Traenkner JJ, Ponce PO, Patterson JE, Goepfert PA, Sofarelli TA, Mocherla S, Ko ER, Ponce de Leon A, Doernberg SB, Atmar RL, Maves RC, Dangond F, Ferreira J, Green M, Makowski M, Bonnett T, Beresnev T, Ghazaryan V, Dempsey W, Nayak SU, Dodd L, Tomashek KM, Beigel JH; ACTT-3 study group members. Efficacy of interferon beta-1a plus remdesivir compared with remdesivir alone in hospitalised adults with COVID-19: a double-bind, randomised, placebo-controlled, phase 3 trial. Lancet Respir Med. 2021 Dec;9(12):1365-1376. doi: 10.1016/S2213-2600(21)00384-2. Epub 2021 Oct 18. PMID 34672949
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343
- [Derived] Azzi Y, Bartash R, Scalea J, Loarte-Campos P, Akalin E. COVID-19 and Solid Organ Transplantation: A Review Article. Transplantation. 2021 Jan 1;105(1):37-55. doi: 10.1097/TP.0000000000003523. PMID 33148977

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the participating sites from those admitted with symptoms of COVID-19 confirmed by PCR. Enrollment occurred between 05AUG2020 and 11NOV2020.
Period: Overall Study
Arm/Group | Remdesivir Plus Interferon Beta-1a | Remdesivir Plus Placebo
Started | 487 | 482
ITT and Modified ITT Population | 487 | 482
As Treated Population | 477 | 468
Completed | 473 | 474
Not Completed | 14 | 8
Not completed — Enrolled but not treated | 8 | 8
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Became ineligible after enrollment | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Remdesivir Plus Interferon Beta-1a | Remdesivir Plus Placebo | Total
Number analyzed (Participants) | 487 | 482 | 969
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 301 | 304 | 605
  >=65 years | 186 | 178 | 364
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (15.8) | 59.1 (16.1) | 58.7 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 190 | 216 | 406
  Male | 297 | 266 | 563
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 154 | 157 | 311
  Not Hispanic or Latino | 323 | 317 | 640
  Unknown or Not Reported | 10 | 8 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 3 | 11
  Asian | 44 | 39 | 83
  Native Hawaiian or Other Pacific Islander | 4 | 5 | 9
  Black or African American | 76 | 84 | 160
  White | 299 | 285 | 584
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 54 | 63 | 117
Region of Enrollment [Number; unit: participants]
  South Korea | 16 | 14 | 30
  Singapore | 3 | 2 | 5
  United States | 432 | 428 | 860
  Japan | 8 | 9 | 17
  Mexico | 28 | 29 | 57
Baseline Ordinal Score [Count of Participants; unit: Participants] — Participants were scored at baseline based on their hospitalization and oxygen usage with enrollment limited to scores 4-6. Ordinal Score 4: Hospitalized, not requiring supplemental oxygen. Ordinal Score 5: Hospitalized, requiring supplemental oxygen. Ordinal Score 6: Hospitalized, on non-invasive ventilation or high flow oxygen devices.
  Participants
    Ordinal Score 4 | 84 | 68 | 152
    Ordinal Score 5 | 368 | 380 | 748
    Ordinal Score 6 | 35 | 34 | 69

OUTCOME MEASURES:

1. Primary Outcome: Time to Recovery for Participants With Baseline Ordinal Score 4, 5 and 6
Description: Day of recovery is defined as the first day on which the subject satisfies one of the following three categories from the ordinal scale: 1) Not hospitalized, no limitations on activities; 2) Not hospitalized, but new or increased limitation on activities and/or new or increased requirement for home oxygen; 3) Hospitalized, not requiring supplemental oxygen and no longer requires ongoing medical care.
Time Frame: Day 1 through Day 29
Population: The modified intention-to-treat (mITT) population includes all participants who were randomized. mITT participants were classified by their randomized treatment assignment and their baseline ordinal score, which is not necessarily equivalent to the disease severity stratum to which the participant was randomized at enrollment.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Remdesivir Plus Interferon Beta-1a | Remdesivir Plus Placebo
Number analyzed (Participants) | 487 | 482
Days | 5.0 [NA to NA] — A large number of participants at the median estimate means there is little variability at the 50th percentile and the methodology described by Klein and Moeschberger (1997) is unable to compute a confidence interval. Also, if less than 50% of participants recover then the median time can not be estimated. | 5.0 [NA to NA] — A large number of participants at the median estimate means there is little variability at the 50th percentile and the methodology described by Klein and Moeschberger (1997) is unable to compute a confidence interval. Also, if less than 50% of participants recover then the median time can not be estimated.
Statistical Analysis 1: Comparison: Remdesivir Plus Interferon Beta-1a vs Remdesivir Plus Placebo; Test type: Superiority; p = 0.880, Log Rank; Cox Proportional Hazard = 0.99, 95% CI 2-sided [0.87 to 1.13]

2. Secondary Outcome: Change From Baseline in Alanine Aminotransferase (ALT)
Description: Blood to evaluate ALT was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge. The measure was assessed by baseline ordinal scale category (categories 4 and 5 versus category 6).
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: The safety population includes all treated participants with available data at baseline and the post baseline assessment point, analyzed as treated.
Measure: Mean (95% Confidence Interval); unit: Units/Liter (U/L)
Groups:
- Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5: 200 mg of Remdesivir administered intravenously on Day 1, followed by a 100 mg once-daily maintenance dose of Remdesivir while hospitalized for up to a 10-day total course and 44 mcg of interferon beta-1a administered by a 0.5 mL subcutaneous injection on Days 1, 3, 5, and 7 while hospitalized for a total of 4 doses in participants with a Baseline Ordinal Score of 4 and 5.
- Remdesivir Plus Interferon Beta-1a in Ordinal Score 6: 200 mg of Remdesivir administered intravenously on Day 1, followed by a 100 mg once-daily maintenance dose of Remdesivir while hospitalized for up to a 10-day total course and 44 mcg of interferon beta-1a administered by a 0.5 mL subcutaneous injection on Days 1, 3, 5, and 7 while hospitalized for a total of 4 doses in participants with a Baseline Ordinal Score of 6
- Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5: 200 mg of Remdesivir administered intravenously on Day 1, followed by a 100 mg once-daily maintenance dose of Remdesivir while hospitalized for up to a 10-day total course and a 0.5 mL placebo injection administered subcutaneously on Days 1, 3, 5, and 7 while hospitalized for a total of 4 doses in participants with a Baseline Ordinal Score of 4 and 5.
- Remdesivir Plus Placebo in Baseline Ordinal Score 6: 200 mg of Remdesivir administered intravenously on Day 1, followed by a 100 mg once-daily maintenance dose of Remdesivir while hospitalized for up to a 10-day total course and a 0.5 mL placebo injection administered subcutaneously on Days 1, 3, 5, and 7 while hospitalized for a total of 4 doses in participants with a Baseline Ordinal Score of 6.
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 6
Number analyzed (Participants) | 432 | 34 | 418 | 31
Units/Liter (U/L)
  Day 3 | 17.6 [13.7 to 21.5] | 2.6 [-4.6 to 9.8] | 5.0 [2.1 to 7.9] | 10.9 [-11.9 to 33.6]
  Day 5: number analyzed (Participants) | 312 | 32 | 291 | 31
  Day 5 | 41.4 [32.7 to 50.0] | 1.5 [-8.5 to 11.5] | 13.5 [9.0 to 18.0] | 3.8 [-9.9 to 17.4]
  Day 8: number analyzed (Participants) | 145 | 29 | 139 | 21
  Day 8 | 18.8 [10.4 to 27.3] | 4.0 [-8.6 to 16.6] | 5.3 [0.0 to 10.6] | -8.7 [-23.4 to 6.0]
  Day 11: number analyzed (Participants) | 72 | 22 | 94 | 16
  Day 11 | 9.9 [-0.6 to 20.4] | -15.1 [-27.4 to -2.9] | 9.0 [1.1 to 16.8] | -11.1 [-28.1 to 5.8]
  Day 15: number analyzed (Participants) | 180 | 21 | 180 | 13
  Day 15 | 3.5 [-2.0 to 9.0] | -4.9 [-19.5 to 9.7] | 2.6 [-2.1 to 7.4] | -17.6 [-43.7 to 8.4]
  Day 29: number analyzed (Participants) | 191 | 10 | 179 | 6
  Day 29 | -3.2 [-13.9 to 7.5] | -9.3 [-54.1 to 35.5] | -6.4 [-13.3 to 0.6] | -13.8 [-51.5 to 23.8]

3. Secondary Outcome: Change From Baseline in Aspartate Aminotransferase (AST)
Description: Blood to evaluate AST was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge. The measure was assessed by baseline ordinal scale category (categories 4 and 5 versus category 6).
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: U/L
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 6
Number analyzed (Participants) | 429 | 34 | 416 | 31
U/L
  Day 3 | 8.0 [4.7 to 11.4] | -5.1 [-15.8 to 5.5] | -4.6 [-8.3 to 0.8] | -10.0 [-23.4 to 3.3]
  Day 5: number analyzed (Participants) | 309 | 32 | 289 | 31
  Day 5 | 13.2 [7.7 to 18.6] | -11.3 [-20.0 to -2.6] | -5.2 [-8.6 to 1.7] | -19.8 [-32.2 to -7.3]
  Day 8: number analyzed (Participants) | 144 | 29 | 139 | 21
  Day 8 | -6.2 [-15.0 to 2.6] | -10.8 [-20.5 to -1.1] | -16.5 [-21.5 to -11.5] | -20.6 [-39.2 to -1.9]
  Day 11: number analyzed (Participants) | 72 | 22 | 94 | 16
  Day 11 | -12.6 [-22.3 to -2.9] | -27.2 [-39.3 to -15.1] | -13.5 [-22.9 to -4.0] | -26.3 [-47.7 to -4.9]
  Day 15: number analyzed (Participants) | 180 | 21 | 179 | 13
  Day 15 | -10.9 [-14.9 to -6.9] | -19.0 [-32.0 to -6.0] | -13.9 [-18.2 to -9.6] | -30.8 [-60.8 to -0.7]
  Day 29: number analyzed (Participants) | 191 | 10 | 179 | 6
  Day 29 | -10.8 [-16.3 to -5.3] | -26.3 [-58.0 to 5.4] | -15.8 [-23.3 to -8.2] | -22.2 [-50.7 to 6.4]

4. Secondary Outcome: Change From Baseline in C-reactive Protein (CRP)
Description: Blood to evaluate CRP was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge. The measure was assessed by baseline ordinal scale category (categories 4 and 5 versus category 6).
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: The mITT population includes all participants by their randomized treatment assignment and baseline ordinal score. For any missing data, if results were available for visits before or after that visit, the average of the two nearest visits was imputed for all missing visits between them. If a subject died or was lost to follow-up, their last available observation was carried forward. If baseline was missing, another pre-treatment dose was used, or the earliest post-treatment dose was used.
  .
Measure: Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 6
Number analyzed (Participants) | 432 | 34 | 429 | 31
mg/L
  Day 3 | -44.3 [-52.4 to -36.2] | -46.6 [-73.0 to -20.3] | -40.0 [-45.9 to -34.0] | -37.6 [-68.8 to -6.3]
  Day 5 | -59.0 [-69.2 to -48.7] | -55.6 [-87.0 to -24.1] | -58.2 [-67.0 to -49.4] | -40.5 [-76.7 to -4.3]
  Day 8 | -63.8 [-72.6 to -55.0] | -57.4 [-96.3 to -18.6] | -63.3 [-72.7 to -53.9] | -69.3 [-104.8 to -33.9]
  Day 11 | -65.6 [-75.3 to -56.0] | -36.0 [-69.6 to -2.5] | -66.6 [-76.3 to -56.9] | -75.6 [-107.0 to -44.2]
  Day 15 | -66.6 [-76.4 to -56.8] | -27.8 [-71.6 to 16.0] | -65.6 [-75.4 to -55.7] | -72.1 [-106.0 to -38.1]
  Day 29 | -69.2 [-79.6 to -58.8] | -46.5 [-91.8 to -1.2] | -70.2 [-81.3 to -59.2] | -76.8 [-110.0 to -43.6]

5. Secondary Outcome: Change From Baseline in Creatinine
Description: Blood to evaluate serum creatinine was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge. The measure was assessed by baseline ordinal scale category (categories 4 and 5 versus category 6).
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 6
Number analyzed (Participants) | 431 | 34 | 420 | 31
mg/dL
  Day 3 | -0.076 [-0.098 to -0.054] | 0.054 [-0.242 to 0.349] | -0.069 [-0.102 to -0.036] | -0.074 [-0.169 to 0.021]
  Day 5: number analyzed (Participants) | 311 | 32 | 292 | 31
  Day 5 | -0.122 [-0.160 to -0.084] | 0.121 [-0.219 to 0.461] | -0.077 [-0.109 to -0.046] | -0.050 [-0.174 to 0.074]
  Day 8: number analyzed (Participants) | 146 | 29 | 139 | 21
  Day 8 | -0.144 [-0.209 to -0.078] | 0.415 [-0.261 to 1.091] | -0.109 [-0.195 to -0.023] | 0.005 [-0.141 to 0.151]
  Day 11: number analyzed (Participants) | 75 | 22 | 94 | 16
  Day 11 | -0.205 [-0.315 to -0.095] | 0.361 [-0.359 to 1.081] | -0.103 [-0.168 to -0.038] | -0.004 [-0.170 to 0.162]
  Day 15: number analyzed (Participants) | 180 | 21 | 181 | 13
  Day 15 | -0.049 [-0.101 to -0.003] | 0.099 [-0.229 to 0.427] | -0.057 [-0.095 to -0.020] | 0.178 [-0.278 to 0.633]
  Day 29: number analyzed (Participants) | 194 | 10 | 179 | 6
  Day 29 | -0.075 [-0.161 to 0.011] | -0.182 [-0.307 to -0.057] | -0.029 [-0.070 to -0.012] | 0.140 [-0.683 to 0.963]

6. Secondary Outcome: Change From Baseline in D-dimer Concentration
Description: Blood to evaluate d-dimer concentration was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15, and 29
Population: The mITT population includes all participants by their randomized treatment assignment and baseline ordinal score. For any missing data, if results were available for visits before or after that visit, the average of the two nearest visits was imputed for all missing visits between them. If a subject died or was lost to follow-up, their last available observation was carried forward. If baseline was missing, another pre-treatment dose was used, or the earliest post-treatment dose was used.
Measure: Mean (95% Confidence Interval); unit: mg/L fibrinogen-equivalent units (FEU)
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 6
Number analyzed (Participants) | 421 | 35 | 422 | 30
mg/L fibrinogen-equivalent units (FEU)
  Day 3 | -0.2 [-0.4 to 0.1] | 2.2 [-10.4 to 14.9] | 0.1 [-0.3 to 0.4] | 0.5 [-0.5 to 1.4]
  Day 5 | -0.2 [-0.5 to 0.1] | -4.0 [-19.6 to 11.7] | 0.2 [-0.2 to 0.7] | 0.8 [-0.8 to 2.5]
  Day 8 | -0.2 [-0.5 to 0.1] | -9.9 [-23.4 to 3.7] | 0.2 [-0.2 to 0.6] | 0.0 [-1.0 to 0.9]
  Day 11 | -0.2 [-0.5 to 0.1] | -10.9 [-24.5 to 2.8] | 0.1 [-0.3 to 0.4] | -0.3 [-1.2 to 0.7]
  Day 15 | -0.2 [-0.5 to 0.2] | -9.1 [-23.1 to 4.8] | -0.1 [-0.4 to 0.3] | -0.3 [-1.2 to 0.5]
  Day 29 | -0.1 [-0.5 to 0.2] | -8.9 [-23.2 to 5.4] | 0.1 [-0.4 to 0.6] | -0.4 [-1.3 to 0.4]

7. Secondary Outcome: Change From Baseline in Hemoglobin
Description: Blood to evaluate hemoglobin was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge. The outcome was assessed by baseline ordinal scale category (categories 4 and 5 versus category 6).
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: grams/deciliter (g/dL)
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 6
Number analyzed (Participants) | 430 | 34 | 418 | 31
grams/deciliter (g/dL)
  Day 3 | -0.19 [-0.28 to -0.10] | -0.14 [-0.49 to 0.22] | -0.20 [-0.29 to -0.10] | -0.10 [-1.10 to 0.90]
  Day 5: number analyzed (Participants) | 310 | 32 | 292 | 31
  Day 5 | -0.04 [-0.17 to 0.09] | -0.47 [-0.90 to -0.04] | -0.13 [-0.27 to 0.00] | -0.81 [-1.19 to -0.44]
  Day 8: number analyzed (Participants) | 145 | 29 | 138 | 21
  Day 8 | -0.34 [-0.57 to -0.11] | -1.13 [-1.70 to -0.57] | -0.29 [-0.50 to -0.08] | -1.01 [-1.49 to -0.53]
  Day 11: number analyzed (Participants) | 75 | 22 | 94 | 15
  Day 11 | -0.71 [-1.08 to -0.33] | -1.98 [-2.87 to -1.09] | -0.47 [-0.79 to -0.15] | -1.32 [-2.27 to -0.37]
  Day 15: number analyzed (Participants) | 178 | 21 | 179 | 13
  Day 15 | -0.58 [-0.81 to -0.36] | -3.18 [-4.22 to -2.13] | -0.43 [-0.68 to -0.18] | -2.65 [-3.87 to -1.44]
  Day 29: number analyzed (Participants) | 193 | 10 | 175 | 6
  Day 29 | -0.39 [-0.60 to -0.17] | -3.89 [-5.55 to -2.23] | -0.13 [-0.37 to 0.11] | -1.15 [-5.12 to 2.82]

8. Secondary Outcome: Change From Baseline in Prothrombin International Normalized Ratio (INR)
Description: Blood to evaluate INR was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge. The outcome was assessed by baseline ordinal scale category (categories 4 and 5 versus category 6).
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 6
Number analyzed (Participants) | 386 | 30 | 376 | 28
ratio
  Day 3 | -0.03 [-0.09 to 0.03] | 0.05 [0.01 to 0.09] | 0.07 [0.01 to 0.14] | -0.08 [-0.31 to 0.16]
  Day 5: number analyzed (Participants) | 269 | 28 | 268 | 28
  Day 5 | -0.03 [-0.11 to 0.04] | 0.02 [-0.03 to 0.07] | 0.09 [0.04 to 0.15] | -0.08 [-0.32 to 0.16]
  Day 8: number analyzed (Participants) | 130 | 25 | 125 | 19
  Day 8 | -0.07 [-0.19 to 0.05] | 0.01 [-0.06 to 0.09] | 0.04 [-0.09 to 0.17] | 0.02 [-0.06 to 0.09]
  Day 11: number analyzed (Participants) | 63 | 18 | 87 | 13
  Day 11 | 0.05 [-0.14 to 0.24] | 0.02 [-0.07 to 0.12] | 0.06 [-0.01 to 0.13] | 0.05 [-0.07 to 0.16]
  Day 15: number analyzed (Participants) | 166 | 18 | 170 | 12
  Day 15 | -0.09 [-0.17 to -0.01] | 0.02 [-0.07 to 0.12] | -0.09 [-0.18 to 0.00] | 0.01 [-0.16 to 0.18]
  Day 29: number analyzed (Participants) | 174 | 7 | 162 | 6
  Day 29 | -0.07 [-0.13 to 0.00] | 0.00 [-0.22 to 0.22] | -0.10 [-0.20 to 0.00] | -0.11 [-0.31 to 0.09]

9. Secondary Outcome: Change From Baseline in Platelets
Description: Blood to evaluate platelets was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge. The outcome was assessed overall and by baseline ordinal scale category (categories 4 and 5 versus category 6).
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: 10^9 cells/liter
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 6
Number analyzed (Participants) | 430 | 34 | 417 | 31
10^9 cells/liter
  Day 3 | 46.5 [41.7 to 51.2] | 38.4 [12.7 to 64.2] | 57.6 [52.7 to 62.4] | 58.8 [40.2 to 77.5]
  Day 5: number analyzed (Participants) | 310 | 32 | 292 | 31
  Day 5 | 82.1 [73.7 to 90.5] | 63.9 [29.7 to 98.1] | 97.8 [89.6 to 106.0] | 82.2 [52.6 to 111.7]
  Day 8: number analyzed (Participants) | 145 | 29 | 137 | 21
  Day 8 | 96.8 [77.6 to 116.0] | 45.2 [2.2 to 88.3] | 126.8 [110.4 to 143.2] | 92.0 [44.1 to 140.0]
  Day 11: number analyzed (Participants) | 75 | 22 | 94 | 15
  Day 11 | 70.9 [48.2 to 93.6] | 20.0 [-37.4 to 77.5] | 98.9 [78.9 to 118.8] | 61.2 [16.3 to 106.1]
  Day 15: number analyzed (Participants) | 177 | 21 | 179 | 13
  Day 15 | 29.4 [11.6 to 47.2] | -40.0 [-103.0 to 23.0] | 33.3 [18.3 to 48.2] | -14.5 [-66.3 to 37.4]
  Day 29: number analyzed (Participants) | 192 | 10 | 175 | 6
  Day 29 | 56.7 [43.0 to 70.4] | 52.4 [-72.0 to 176.8] | 52.3 [38.5 to 66.1] | 4.5 [-95.6 to 104.6]

10. Secondary Outcome: Change From Baseline in Total Bilirubin
Description: Blood to evaluate total bilirubin was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge. The outcome was assessed by baseline ordinal scale category (categories 4 and 5 versus category 6).
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 6
Number analyzed (Participants) | 429 | 34 | 418 | 31
mg/dL
  Day 3 | -0.08 [-0.10 to -0.06] | 0.07 [-0.02 to 0.17] | -0.07 [-0.09 to -0.05] | 0.03 [-0.05 to 0.11]
  Day 5: number analyzed (Participants) | 310 | 31 | 291 | 31
  Day 5 | -0.07 [-0.10 to -0.03] | 0.03 [-0.05 to 0.11] | 0.00 [-0.04 to 0.03] | 0.02 [-0.07 to 0.11]
  Day 8: number analyzed (Participants) | 145 | 28 | 139 | 21
  Day 8 | -0.03 [-0.09 to 0.02] | 0.10 [0.02 to 0.19] | 0.04 [-0.01 to 0.09] | 0.04 [-0.03 to 0.12]
  Day 11: number analyzed (Participants) | 71 | 22 | 94 | 16
  Day 11 | 0.00 [-0.08 to 0.09] | 0.16 [-0.01 to 0.34] | 0.09 [0.01 to 0.17] | -0.01 [-0.14 to 0.11]
  Day 15: number analyzed (Participants) | 180 | 21 | 180 | 13
  Day 15 | 0.09 [0.02 to 0.15] | 0.34 [0.03 to 0.65] | 0.03 [-0.01 to 0.08] | 0.13 [-0.22 to 0.47]
  Day 29: number analyzed (Participants) | 190 | 10 | 179 | 6
  Day 29 | -0.01 [-0.05 to 0.03] | 0.01 [-0.30 to 0.32] | -0.06 [-0.11 to -0.01] | 0.03 [-0.21 to 0.28]

11. Secondary Outcome: Change From Baseline in White Blood Cell Count (WBC)
Description: Blood to evaluate WBC was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge. The outcome was assessed by baseline ordinal scale category (categories 4 and 5 versus category 6).
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: 10^9 cells/liter
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 6
Number analyzed (Participants) | 430 | 34 | 418 | 31
10^9 cells/liter
  Day 3 | -0.166 [-0.437 to 0.106] | 0.255 [-0.823 to 1.333] | 0.720 [0.446 to 0.994] | 0.856 [-0.800 to 2.512]
  Day 5: number analyzed (Participants) | 310 | 32 | 292 | 31
  Day 5 | 0.486 [0.109 to 0.863] | 0.434 [-0.970 to 1.839] | 1.894 [1.496 to 2.293] | 0.908 [-1.047 to 2.864]
  Day 8: number analyzed (Participants) | 145 | 29 | 138 | 21
  Day 8 | 1.037 [0.449 to 1.626] | 3.062 [1.010 to 5.115] | 3.529 [2.834 to 4.224] | 3.261 [0.890 to 5.632]
  Day 11: number analyzed (Participants) | 75 | 22 | 94 | 15
  Day 11 | 3.145 [1.878 to 4.411] | 4.420 [1.436 to 7.404] | 3.646 [2.659 to 4.632] | 3.153 [0.065 to 6.240]
  Day 15: number analyzed (Participants) | 178 | 21 | 179 | 13
  Day 15 | 0.649 [-0.015 to 1.314] | 3.030 [-0.186 to 6.246] | 1.211 [0.592 to 1.830] | 1.562 [-1.396 to 4.519]
  Day 29: number analyzed (Participants) | 193 | 10 | 175 | 6
  Day 29 | -0.470 [-1.157 to 0.217] | -0.472 [-4.070 to 3.126] | -0.294 [-0.890 to 0.302] | -2.123 [-7.210 to 2.963]

12. Secondary Outcome: Change From Baseline in Neutrophils
Description: Blood to evaluate neutrophils was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge. The outcome was assessed by baseline ordinal scale category (categories 4 and 5 versus category 6).
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: 10^9 cells/liter
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 6
Number analyzed (Participants) | 421 | 33 | 408 | 31
10^9 cells/liter
  Day 3 | -0.622 [-0.880 to -0.365] | -0.324 [-1.346 to 0.698] | 0.329 [0.062 to 0.596] | 0.479 [-1.022 to 1.981]
  Day 5: number analyzed (Participants) | 303 | 31 | 286 | 30
  Day 5 | -0.307 [-0.678 to 0.064] | -0.123 [-1.439 to 1.192] | 1.096 [0.702 to 1.489] | 0.323 [-1.437 to 2.083]
  Day 8: number analyzed (Participants) | 143 | 27 | 134 | 21
  Day 8 | 0.187 [-0.401 to 0.776] | 1.712 [0.108 to 3.316] | 2.583 [1.913 to 3.252] | 2.312 [0.090 to 4.534]
  Day 11: number analyzed (Participants) | 71 | 20 | 90 | 15
  Day 11 | 2.069 [0.770 to 3.368] | 3.419 [0.837 to 6.002] | 2.612 [1.634 to 3.590] | 1.146 [-1.269 to 3.561]
  Day 15: number analyzed (Participants) | 176 | 19 | 178 | 13
  Day 15 | -0.383 [-1.018 to 0.251] | 1.311 [-1.617 to 4.238] | 0.165 [-0.429 to 0.758] | -0.004 [-2.582 to 2.574]
  Day 29: number analyzed (Participants) | 191 | 10 | 175 | 6
  Day 29 | -1.779 [-2.387 to -1.171] | -1.867 [-5.061 to 1.327] | -1.492 [-2.053 to -0.930] | -3.317 [-7.447 to 0.814]

13. Secondary Outcome: Change From Baseline in Lymphoctyes
Description: Blood to evaluate lymphocytes was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge. The outcome was assessed by baseline ordinal scale category (categories 4 and 5 versus category 6).
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: 10^9 cells/liter
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 6
Number analyzed (Participants) | 421 | 33 | 408 | 31
10^9 cells/liter
  Day 3 | 0.301 [0.250 to 0.352] | 0.237 [0.058 to 0.416] | 0.227 [0.128 to 0.326] | 0.137 [-0.004 to 0.277]
  Day 5: number analyzed (Participants) | 303 | 31 | 286 | 30
  Day 5 | 0.492 [0.417 to 0.568] | 0.289 [0.093 to 0.484] | 0.470 [0.392 to 0.548] | 0.242 [0.009 to 0.475]
  Day 8: number analyzed (Participants) | 143 | 27 | 135 | 21
  Day 8 | 0.390 [0.297 to 0.484] | 0.281 [0.104 to 0.458] | 0.404 [0.263 to 0.544] | 0.377 [0.101 to 0.653]
  Day 11: number analyzed (Participants) | 71 | 20 | 90 | 15
  Day 11 | 0.536 [0.352 to 0.719] | 0.347 [0.146 to 0.548] | 0.486 [0.356 to 0.617] | 0.867 [0.186 to 1.547]
  Day 15: number analyzed (Participants) | 177 | 19 | 178 | 13
  Day 15 | 0.655 [0.558 to 0.753] | 0.384 [0.131 to 0.637] | 0.679 [0.557 to 0.801] | 0.642 [0.223 to 1.061]
  Day 29: number analyzed (Participants) | 191 | 10 | 175 | 6
  Day 29 | 0.863 [0.773 to 0.953] | 0.575 [0.264 to 0.885] | 0.909 [0.823 to 0.994] | 0.873 [0.535 to 1.211]

14. Secondary Outcome: Change From Baseline in Monocytes
Description: Blood to evaluate monocytes was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge. The outcome was assessed by baseline ordinal scale category (categories 4 and 5 versus category 6).
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: 10^9 cells/liter
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 6
Number analyzed (Participants) | 420 | 33 | 407 | 31
10^9 cells/liter
  Day 3 | 0.157 [0.131 to 0.184] | 0.112 [0.010 to 0.215] | 0.127 [0.099 to 0.155] | 0.179 [0.040 to 0.318]
  Day 5: number analyzed (Participants) | 303 | 31 | 285 | 30
  Day 5 | 0.229 [0.193 to 0.266] | 0.136 [-0.006 to 0.277] | 0.212 [0.173 to 0.252] | 0.172 [-0.019 to 0.362]
  Day 8: number analyzed (Participants) | 143 | 27 | 134 | 21
  Day 8 | 0.301 [0.244 to 0.359] | 0.147 [0.021 to 0.273] | 0.311 [0.229 to 0.392] | 0.348 [0.155 to 0.541]
  Day 11: number analyzed (Participants) | 71 | 20 | 90 | 15
  Day 11 | 0.381 [0.262 to 0.500] | 0.365 [0.144 to 0.585] | 0.403 [0.303 to 0.503] | 0.333 [-0.022 to 0.689]
  Day 15: number analyzed (Participants) | 177 | 19 | 178 | 13
  Day 15 | 0.207 [0.152 to 0.262] | 0.107 [-0.047 to 0.260] | 0.212 [0.143 to 0.280] | 0.262 [0.077 to 0.447]
  Day 29: number analyzed (Participants) | 191 | 10 | 175 | 6
  Day 29 | 0.131 [0.085 to 0.176] | 0.310 [0.057 to 0.563] | 0.114 [0.069 to 0.160] | 0.015 [-0.807 to 0.838]

15. Secondary Outcome: Change From Baseline in Basophils
Description: Blood to evaluate basophils was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge. The outcome was assessed by baseline ordinal scale category (categories 4 and 5 versus category 6).
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: 10^9 cells/liter
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 6
Number analyzed (Participants) | 417 | 33 | 405 | 30
10^9 cells/liter
  Day 3 | 0.000 [-0.004 to 0.003] | 0.003 [-0.003 to 0.008] | 0.001 [-0.002 to 0.005] | 0.002 [-0.014 to 0.018]
  Day 5: number analyzed (Participants) | 301 | 31 | 284 | 29
  Day 5 | 0.002 [-0.002 to 0.006] | 0.011 [0.001 to 0.021] | 0.009 [0.001 to 0.018] | 0.003 [-0.008 to 0.015]
  Day 8: number analyzed (Participants) | 143 | 27 | 134 | 20
  Day 8 | 0.015 [0.000 to 0.030] | 0.004 [-0.004 to 0.012] | 0.010 [0.001 to 0.018] | 0.007 [-0.001 to 0.014]
  Day 11: number analyzed (Participants) | 70 | 20 | 90 | 15
  Day 11 | 0.009 [0.000 to 0.019] | 0.022 [0.000 to 0.044] | 0.016 [0.009 to 0.023] | 0.015 [0.006 to 0.024]
  Day 15: number analyzed (Participants) | 176 | 19 | 178 | 13
  Day 15 | 0.021 [0.014 to 0.028] | 0.007 [-0.004 to 0.018] | 0.027 [0.021 to 0.034] | 0.022 [0.004 to 0.039]
  Day 29: number analyzed (Participants) | 190 | 10 | 175 | 5
  Day 29 | 0.027 [0.019 to 0.035] | 0.049 [0.013 to 0.085] | 0.031 [0.024 to 0.039] | 0.028 [-0.017 to 0.074]

16. Secondary Outcome: Change From Baseline in Eosinophils
Description: Blood to evaluate eosinophils was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge. The outcome was assessed by baseline ordinal scale category (categories 4 and 5 versus category 6).
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: 10^9 cells/liter
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 6
Number analyzed (Participants) | 417 | 33 | 405 | 30
10^9 cells/liter
  Day 3 | 0.011 [0.002 to 0.019] | 0.014 [-0.001 to 0.029] | 0.013 [0.007 to 0.019] | 0.006 [-0.009 to 0.020]
  Day 5: number analyzed (Participants) | 301 | 31 | 284 | 29
  Day 5 | 0.016 [0.009 to 0.024] | 0.037 [0.009 to 0.066] | 0.032 [0.021 to 0.043] | 0.019 [0.000 to 0.038]
  Day 8: number analyzed (Participants) | 143 | 27 | 134 | 21
  Day 8 | 0.043 [0.031 to 0.054] | 0.028 [0.003 to 0.053] | 0.041 [0.025 to 0.057] | 0.038 [0.001 to 0.074]
  Day 11: number analyzed (Participants) | 71 | 20 | 90 | 15
  Day 11 | 0.044 [0.030 to 0.058] | 0.117 [-0.021 to 0.254] | 0.063 [0.044 to 0.082] | 0.105 [0.058 to 0.151]
  Day 15: number analyzed (Participants) | 176 | 19 | 178 | 13
  Day 15 | 0.116 [0.101 to 0.132] | 0.135 [0.076 to 0.194] | 0.130 [0.112 to 0.147] | 0.166 [0.096 to 0.235]
  Day 29: number analyzed (Participants) | 190 | 10 | 175 | 5
  Day 29 | 0.189 [0.135 to 0.243] | 0.291 [0.060 to 0.521] | 0.172 [0.152 to 0.192] | 0.199 [0.025 to 0.374]

17. Secondary Outcome: Change in National Early Warning Score (NEWS) From Baseline
Description: The NEW score has demonstrated an ability to discriminate patients at risk of poor outcomes. This score is based on 7 clinical parameters (respiration rate, oxygen saturation, any supplemental oxygen, temperature, systolic blood pressure, heart rate, level of consciousness). The NEW Score is being used as an efficacy measure. The minimum score is 0, representing the better outcome, and the maximum value is 19, representing the worse outcome.
Time Frame: Days 1, 3, 5, 8, 11, 15, 22, and 29
Population: The intent-to-treat (ITT) population includes all participants who were randomized with data at baseline and at each timepoint. Missing values were imputed using Last Observation Carried Forward.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 6
Number analyzed (Participants) | 452 | 35 | 448 | 34
units on a scale
  Day 3 | -0.7 [-0.9 to -0.5] | 1.0 [0.0 to 2.0] | -0.6 [-0.8 to -0.4] | -0.7 [-1.7 to 0.3]
  Day 5 | -1.1 [-1.3 to -0.8] | 1.6 [0.4 to 2.8] | -1.0 [-1.2 to -0.7] | -1.3 [-2.3 to -0.3]
  Day 8 | -1.4 [-1.6 to -1.1] | 1.7 [0.3 to 3.2] | -1.3 [-1.5 to -1.0] | -0.6 [-2.2 to 0.9]
  Day 11 | -1.6 [-1.8 to -1.3] | 1.4 [-0.2 to 3.0] | -1.4 [-1.7 to -1.2] | -1.0 [-2.7 to 0.7]
  Day 15 | -1.6 [-1.9 to -1.4] | 1.9 [0.0 to 3.7] | -1.6 [-1.9 to -1.2] | -1.5 [-3.2 to 0.2]
  Day 22 | -1.5 [-1.8 to -1.2] | 1.6 [-0.5 to 3.8] | -1.6 [-2.0 to -1.3] | -1.7 [-3.8 to 0.4]
  Day 29 | -1.7 [-2.1 to -1.4] | 1.9 [-0.4 to 4.3] | -1.9 [-2.2 to -1.5] | -1.8 [-3.9 to 0.3]

18. Secondary Outcome: Percentage of Participants Reporting Grade 3 and 4 Clinical and/or Laboratory Adverse Events (AEs)
Description: Grade 3 AEs are defined as events that interrupt usual activities of daily living, or significantly affects clinical status, or may require intensive therapeutic intervention. Severe events are usually incapacitating. Grade 4 AEs are defined as events that are potentially life threatening.
Time Frame: Day 1 through Day 29
Population: The safety population includes all participants with available data post baseline, analyzed as treated.
Measure: Number; unit: percentage of participants
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 6
Number analyzed (Participants) | 442 | 35 | 435 | 33
percentage of participants | 38.9 | 60.0 | 31.7 | 36.4
Statistical Analysis 1: Comparison: Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 vs Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5; Test type: Superiority; Risk Difference (RD) = 7.2, 95% CI 2-sided [0.9 to 13.4]
Statistical Analysis 2: Comparison: Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 vs Remdesivir Plus Placebo in Baseline Ordinal Score 6; Test type: Superiority; Risk Difference (RD) = 23.6, 95% CI 2-sided [0.0 to 43.9]

19. Secondary Outcome: Percentage of Participants Reporting Serious Adverse Events (SAEs)
Description: An SAE is defined as an AE or suspected adverse reaction is considered serious if, in the view of either the investigator or the sponsor, it results in death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect.
Time Frame: Day 1 through Day 29
Population: The safety population includes all participants with available data post baseline, analyzed as treated.
Measure: Number; unit: percentage of participants
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 6
Number analyzed (Participants) | 442 | 35 | 435 | 33
percentage of participants | 14.7 | 60.0 | 13.3 | 24.2
Statistical Analysis 1: Comparison: Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 vs Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5; Test type: Superiority; Risk Difference (RD) = 1.4, 95% CI 2-sided [-3.2 to 6.0]
Statistical Analysis 2: Comparison: Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 vs Remdesivir Plus Placebo in Baseline Ordinal Score 6; Test type: Superiority; Risk Difference (RD) = 35.8, 95% CI 2-sided [12.3 to 54.2]

20. Secondary Outcome: Duration of Hospitalization
Description: Duration of hospitalization was determined two ways. The first includes imputations for participants who died. The second method is restricted to participants who did not die.
Time Frame: Day 1 through Day 29
Population: The intent-to-treat (ITT) population includes all participants who were randomized.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 6
Number analyzed (Participants) | 452 | 35 | 448 | 34
Days
  Including imputations for participants who died | 6 [4 to 9] | 28 [9 to 28] | 6 [4 to 10] | 10 [7 to 17]
  Among participants who did not die: number analyzed (Participants) | 438 | 28 | 435 | 30
  Among participants who did not die | 6 [4 to 9] | 16.5 [8.5 to 28] | 6 [4 to 9] | 10 [7 to 14]

21. Secondary Outcome: Duration of Invasive Mechanical Ventilation
Description: Duration of invasive ventilation was measured in days among participants who required invasive ventilation, determined two ways. The first includes imputations for participants who died. The second method is restricted to participants who did not die
Time Frame: Day 1 through Day 29
Population: The analysis population is restricted to randomized participants who were on invasive ventilation.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 6
Number analyzed (Participants) | 20 | 19 | 21 | 5
Days
  Including imputations for participants who died | 28 [15 to 28] | 23 [14 to 28] | 26.5 [12 to 28] | 28 [20 to 28]
  Among participants who did not die: number analyzed (Participants) | 11 | 14 | 15 | 2
  Among participants who did not die | 14 [6 to 16] | 19 [9 to 23] | 14 [7 to 20] | 13.5 [7 to 20]

22. Secondary Outcome: Duration of New Non-invasive Ventilation or High Flow Oxygen Use
Description: Duration of new non-invasive ventilation or high flow oxygen use was measured in days among participants who were not on non-invasive ventilation or high-flow oxygen use at baseline, determined two ways. The first includes imputations for participants who died. The second method is restricted to participants who did not die
Time Frame: Day 1 through Day 29
Population: The analysis population is restricted to randomized participants who were not on noninvasive ventilation or high-flow oxygen at baseline but who subsequently required non-invasive or high-flow oxygen.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5
Number analyzed (Participants) | 67 | 67
Days
  Including imputations for participants who died | 5 [2 to 12] | 6 [3 to 14]
  Among participants who did not die: number analyzed (Participants) | 57 | 57
  Among participants who did not die | 4 [2 to 7] | 5 [3 to 7]

23. Secondary Outcome: Duration of New Oxygen Use
Description: Duration of new oxygen use was measured in days among participants who were not on oxygen at baseline, determined two ways. The first includes imputations for participants who died. The second method is restricted to participants who did not die
Time Frame: Day 1 through Day 29
Population: The analysis population is restricted to randomized participants who were not on oxygen at baseline but who subsequently required oxygen.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5
Number analyzed (Participants) | 43 | 39
Days
  Including imputations for participants who died | 3 [1 to 10] | 3 [1 to 8]
  Among participants who did not die: number analyzed (Participants) | 41 | 39
  Among participants who did not die | 3 [1 to 7] | 3 [1 to 8]

24. Secondary Outcome: Duration of New Ventilator or Extracorporeal Membrane Oxygenation (ECMO) Use
Description: Duration of new ventilator or ECMO use was measured in days among participants who were not on a ventilator or ECMO at baseline, determined two ways. The first includes imputations for participants who died. The second method is restricted to participants who did not die.
Time Frame: Day 1 through Day 29
Population: The analysis population is restricted to randomized participants not on a ventilator or ECMO at baseline but who subsequently required a ventilator or ECMO.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 6
Number analyzed (Participants) | 20 | 19 | 21 | 5
Days
  Including imputations for participants who died | 28 [15 to 28] | 23 [14 to 28] | 26.5 [12 to 28] | 28 [20 to 28]
  Among participants who did not die: number analyzed (Participants) | 11 | 14 | 15 | 2
  Among participants who did not die | 14 [6 to 16] | 19 [9 to 23] | 14 [7 to 20] | 13.5 [7 to 20]

25. Secondary Outcome: Duration of Non Invasive Ventilation or High Flow Oxygen Use
Description: Duration of non invasive ventilation or high flow oxygen use was measured in days, determined two ways. The first includes imputations for participants who died. The second method is restricted to participants who did not die.
Time Frame: Day 1 through Day 29
Population: The analysis population is restricted to participants who required non invasive ventilation or high flow oxygen use.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 6
Number analyzed (Participants) | 67 | 35 | 67 | 34
Days
  Including imputations for participants who died | 5 [2 to 12] | 6 [3 to 28] | 6 [3 to 14] | 5.5 [3 to 10]
  Among participants who did not die: number analyzed (Participants) | 57 | 28 | 57 | 30
  Among participants who did not die | 4 [2 to 7] | 4 [3 to 7] | 5 [3 to 7] | 4 [2 to 7]

26. Secondary Outcome: Duration of Oxygen Use
Description: Duration of oxygen use was measured in days among participants who were on oxygen in based, calculated in two ways. The first includes imputations for participants who died. The second method is restricted to participants who did not die.
Time Frame: Day 1 through Day 29
Population: The analysis population is restricted to randomized participants who were on oxygen at baseline.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 6
Number analyzed (Participants) | 368 | 35 | 380 | 34
Days
  Including imputations for participants who died | 6 [3 to 22.5] | 28 [15 to 28] | 7.5 [3 to 24] | 21.5 [9 to 28]
  Among participants who did not die: number analyzed (Participants) | 356 | 28 | 367 | 30
  Among participants who did not die | 6 [3 to 20.5] | 27.5 [14.5 to 28] | 7 [3 to 23] | 20.5 [9 to 28]

27. Secondary Outcome: Number of Participants With Discontinuation or Temporary Suspension of Study Product Administration
Description: Discontinuation or temporary suspension of study product administration, including participants who died or were discharged, was evaluated by baseline ordinal scale category (categories 4 and 5 versus category 6).
Time Frame: Day 1 through Day 10
Population: The ITT population incudes all participants who were randomized
Measure: Count of Participants; unit: Participants
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 6
Number analyzed (Participants) | 443 | 35 | 441 | 34
Participants
  Remdesivir | 400 | 25 | 382 | 22
  Interferon Beta-1a/Placebo | 337 | 13 | 341 | 19

28. Secondary Outcome: Proportion of Participants With New Non-invasive Ventilation or High Flow Oxygen Use
Description: Proportion of participants with new non-invasive ventilation or high flow oxygen use was assessed as for participants in Ordinal Score 4 and 5.
Time Frame: Day 1 through Day 29
Population: The modified intention-to-treat (mITT) population includes all Ordinal Score 4 and 5 participants who were randomized. mITT participants were classified by their randomized treatment assignment and their baseline ordinal score, which is not necessarily equivalent to the disease severity stratum to which the participant was randomized at enrollment.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5
Number analyzed (Participants) | 452 | 448
Proportion of participants | 0.15 [0.12 to 0.18] | 0.15 [0.12 to 0.19]

29. Secondary Outcome: Proportion of Participants With New Oxygen Use
Description: Incidence of new oxygen use was assessed as for participants in Ordinal Score 4 and 5 who were not on oxygen at baseline.
Time Frame: Day 1 through Day 29
Population: The modified intention-to-treat (mITT) population includes all participants in Ordinal Score 4 and 5 who were randomized and not on oxygen at baseline. mITT participants were classified by their randomized treatment assignment and their baseline ordinal score, which is not necessarily equivalent to the disease severity stratum to which the participant was randomized at enrollment.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5
Number analyzed (Participants) | 84 | 68
Proportion of participants | 0.51 [0.41 to 0.62] | 0.57 [0.46 to 0.68]

30. Secondary Outcome: Proportion of Participants With New Ventilator or Extracorporeal Membrane Oxygenation (ECMO) Use
Description: Incidence of new ventilator or extracorporeal membrane oxygenation (ECMO) use was assessed among participants not on ventilator or extracorporeal membrane oxygenation (ECMO) use at baseline.
Time Frame: Day 1 through Day 29
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 6
Number analyzed (Participants) | 452 | 35 | 448 | 34
Proportion of participants | 0.04 [0.03 to 0.07] | 0.54 [0.38 to 0.70] | 0.05 [0.03 to 0.07] | 0.15 [0.06 to 0.30]

31. Secondary Outcome: Mean Change From Baseline in the Ordinal Scale
Description: The ordinal scale is an assessment of the clinical status at the first assessment of a given study day. The scale is as follows: 1) Not hospitalized, no limitations on activities; 2) Not hospitalized, but new or increased limitation on activities and/or new or increased requirement for home oxygen; 3) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 5) Hospitalized, requiring supplemental oxygen; 6) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 7) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 8) Death. A positive change indicates a worsening and a negative change is an improvement.
Time Frame: Day 1, 3, 5, 8, 11, 15, 22, and 29
Population: The intent-to-treat (ITT) population includes all participants who were randomized reporting a clinical score. Missing values were imputed using Last Observation Carried Forward.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 6
Number analyzed (Participants) | 452 | 35 | 448 | 34
units on a scale
  Day 3 | 0.1 [0.0 to 0.1] | 0.1 [0.0 to 0.3] | 0.1 [0.0 to 0.1] | 0.0 [-0.2 to 0.1]
  Day 5 | -0.1 [-0.1 to 0.0] | 0.3 [0.1 to 0.6] | 0.0 [-0.1 to 0.0] | -0.1 [-0.3 to 0.1]
  Day 8 | -0.2 [-0.3 to -0.1] | 0.3 [-0.1 to 0.6] | -0.1 [-0.2 to 0.0] | -0.4 [-0.8 to 0.0]
  Day 11 | -0.4 [-0.5 to -0.3] | 0.1 [-0.4 to 0.5] | -0.4 [-0.5 to -0.3] | -0.6 [-1.0 to -0.2]
  Day 15 | -2.5 [-2.7 to -2.4] | -0.8 [-1.7 to 0.0] | -2.5 [-2.7 to -2.3] | -2.3 [-3.0 to -1.5]
  Day 22 | -2.8 [-2.9 to -2.6] | -1.3 [-2.3 to -0.4] | -2.8 [-2.9 to -2.7] | -2.9 [-3.7 to -2.1]
  Day 29 | -2.9 [-3.0 to -2.7] | -1.5 [-2.5 to -0.5] | -3.0 [-3.1 to -2.8] | -3.2 [-4.0 to -2.4]

32. Secondary Outcome: Percentage of Participants at Each Clinical Status Using Ordinal Scale at Day 15 for Participants With Baseline Ordinal Score 4 and 5
Description: The ordinal scale is an assessment of the clinical status at the first assessment of a given study day. The scale is as follows: 8) Death; 7) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 6) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 5) Hospitalized, requiring supplemental oxygen; 4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 3) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 2) Not hospitalized, limitation on activities and/or requiring home oxygen; 1) Not hospitalized, no limitations on activities. Data was imputed using last observation carried forward or worst possible score based on hospitalization status (2 if not hospitalized, 7 if hospitalized) when there was a change in hospitalization status since last score. Deaths were imputed as an 8.
Time Frame: Day 15
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5
Number analyzed (Participants) | 452 | 448
percentage of participants
  Death at or before study visit | 1.3 [0.6 to 2.9] | 2.0 [1.1 to 3.8]
  Hospitalized, on invasive mech. vent. or ECMO | 2.2 [1.2 to 4.0] | 3.1 [1.9 to 5.2]
  Hospitalized, on noninvasive vent./high flow O2 | 1.1 [0.5 to 2.6] | 1.8 [0.9 to 3.5]
  Hospitalized, requiring supplemental oxygen | 6.0 [4.1 to 8.6] | 6.0 [4.2 to 8.6]
  Hospitalized, not on O2, requiring ongoing care | 3.1 [1.9 to 5.1] | 2.5 [1.4 to 4.3]
  Hospitalized, not requiring O2, no longer req care | 0.4 [0.1 to 1.6] | 0.9 [0.3 to 2.3]
  Not hospitalized, limit on activities/req home O2 | 53.1 [48.5 to 57.7] | 52.5 [47.8 to 57.0]
  Not hospitalized, no limitations on activities | 32.7 [28.6 to 37.2] | 31.3 [27.1 to 35.7]

33. Secondary Outcome: Percentage of Participants Reporting Each Severity Rating on an 8 Point Ordinal Scale at Day 1
Description: The ordinal scale is an assessment of the clinical status at the first assessment of a given study day. The scale is as follows: 8) Death; 7) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 6) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 5) Hospitalized, requiring supplemental oxygen; 4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 3) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 2) Not hospitalized, limitation on activities and/or requiring home oxygen; 1) Not hospitalized, no limitations on activities.
Time Frame: Day 1
Population: The intent-to-treat (ITT) population includes all participants who were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 6
Number analyzed (Participants) | 452 | 35 | 448 | 34
percentage of participants
  Death at or before study visit | 0.0 [0.0 to 0.8] | 0.0 [0.0 to 9.9] | 0.0 [0.0 to 0.9] | 0.0 [0.0 to 10.2]
  Hospitalized, on invasive mech. vent. or ECMO | 0.0 [0.0 to 0.8] | 0.0 [0.0 to 9.9] | 0.0 [0.0 to 0.9] | 0.0 [0.0 to 10.2]
  Hospitalized, on non-invasive vent./high flow O2 | 81.4 [77.6 to 84.7] | 100 [90.1 to 100] | 84.8 [81.2 to 87.8] | 100 [89.8 to 100.0]
  Hospitalized, requiring supplemental oxygen | 18.6 [15.3 to 22.4] | 0.0 [0.0 to 9.9] | 15.2 [12.2 to 18.8] | 0.0 [0.0 to 10.2]
  Hospitalized, not on O2, requiring ongoing care | 0.0 [0.0 to 0.8] | 0.0 [0.0 to 9.9] | 0.0 [0.0 to 0.9] | 0.0 [0.0 to 10.2]
  Hospitalized, not requiring O2, no longer req care | 0.0 [0.0 to 0.8] | 0.0 [0.0 to 9.9] | 0.0 [0.0 to 0.9] | 0.0 [0.0 to 10.2]
  Not hospitalized, limit on activities/req home O2 | 0.0 [0.0 to 0.8] | 0.0 [0.0 to 9.9] | 0.0 [0.0 to 0.9] | 0.0 [0.0 to 10.2]
  Not hospitalized, no limitations on activities | 0.0 [0.0 to 0.8] | 0.0 [0.0 to 9.9] | 0.0 [0.0 to 0.9] | 0.0 [0.0 to 10.2]

34. Secondary Outcome: Percentage of Participants Reporting Each Severity Rating on an 8 Point Ordinal Scale at Day 3
Description: as for outcome 33
Time Frame: Day 3
Population: The intent-to-treat (ITT) population includes all participants who were randomized. Missing values were imputed using Last Observation Carried Forward.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 6
Number analyzed (Participants) | 452 | 35 | 448 | 34
percentage of participants
  Death at or before study visit | 0.0 [0.0 to 0.8] | 0.0 [0.0 to 9.9] | 0.2 [0.0 to 1.3] | 0.0 [0.0 to 10.2]
  Hospitalized, on invasive mech. vent. or ECMO | 0.9 [0.3 to 2.3] | 17.1 [8.1 to 32.7] | 1.6 [0.8 to 3.2] | 5.9 [1.6 to 19.1]
  Hospitalized, on non-invasive vent./high flow O2 | 6.0 [4.1 to 8.6] | 80.0 [64.1 to 90.0] | 6.3 [4.4 to 8.9] | 85.3 [69.9 to 93.6]
  Hospitalized, requiring supplemental oxygen | 74.1 [69.9 to 77.9] | 2.9 [0.5 to 14.5] | 73.7 [69.4 to 77.5] | 8.8 [3.0 to 23.0]
  Hospitalized, not on O2, requiring ongoing care | 18.8 [15.5 to 22.7] | 0.0 [0.0 to 9.9] | 18.1 [14.8 to 21.9] | 0.0 [0.0 to 10.2]
  Hospitalized, not requiring O2, no longer req care | 0.2 [0.0 to 1.2] | 0.0 [0.0 to 9.9] | 0.0 [0.0 to 0.9] | 0.0 [0.0 to 10.2]
  Not hospitalized, limit on activities/req home O2 | 0.0 [0.0 to 0.8] | 0.0 [0.0 to 9.9] | 0.2 [0.0 to 1.3] | 0.0 [0.0 to 10.2]
  Not hospitalized, no limitations on activities | 0.0 [0.0 to 0.8] | 0.0 [0.0 to 9.9] | 0.0 [0.0 to 0.9] | 0.0 [0.0 to 10.2]

35. Secondary Outcome: Percentage of Participants Reporting Each Severity Rating on an 8 Point Ordinal Scale at Day 5
Description: as for outcome 33
Time Frame: Day 5
Population: as for outcome 34
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 6
Number analyzed (Participants) | 452 | 35 | 448 | 34
percentage of participants
  Death at or before study visit | 0.2 [0.0 to 1.2] | 2.9 [0.5 to 14.5] | 0.7 [0.2 to 2.0] | 0.0 [0.0 to 10.2]
  Hospitalized, on invasive mech. vent. or ECMO | 1.8 [0.9 to 3.5] | 37.1 [23.2 to 53.7] | 2.7 [1.5 to 4.6] | 14.7 [6.4 to 30.1]
  Hospitalized, on non-invasive vent./high flow O2 | 8.4 [6.2 to 11.3] | 48.6 [33.0 to 64.4] | 8.7 [6.4 to 11.7] | 58.8 [42.2 to 73.6]
  Hospitalized, requiring supplemental oxygen | 49.1 [44.5 to 53.7] | 11.4 [4.5 to 26.0] | 46.2 [41.6 to 50.8] | 20.6 [10.3 to 36.8]
  Hospitalized, not on O2, requiring ongoing care | 26.5 [22.7 to 30.8] | 0.0 [0.0 to 9.9] | 26.3 [22.5 to 30.6] | 0.0 [0.0 to 10.2]
  Hospitalized, not requiring O2, no longer req care | 0.7 [0.2 to 1.9] | 0.0 [0.0 to 9.9] | 0.0 [0.0 to 0.9] | 0.0 [0.0 to 10.2]
  Not hospitalized, limit on activities/req home O2 | 13.3 [10.5 to 16.7] | 0.0 [0.0 to 9.9] | 15.2 [12.2 to 18.8] | 5.9 [1.6 to 19.1]
  Not hospitalized, no limitations on activities | 0.0 [0.0 to 0.8] | 0.0 [0.0 to 9.9] | 0.2 [0.0 to 1.3] | 0.0 [0.0 to 10.2]

36. Secondary Outcome: Percentage of Participants Reporting Each Severity Rating on an 8 Point Ordinal Scale at Day 8
Description: as for outcome 33
Time Frame: Day 8
Population: as for outcome 34
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 6
Number analyzed (Participants) | 452 | 35 | 448 | 34
percentage of participants
  Death at or before study visit | 0.2 [0.0 to 1.2] | 5.7 [1.6 to 18.6] | 0.9 [0.3 to 2.3] | 5.9 [1.6 to 19.1]
  Hospitalized, on invasive mech. vent. or ECMO | 2.7 [1.5 to 4.6] | 45.7 [30.5 to 61.8] | 2.9 [1.7 to 4.9] | 11.8 [4.7 to 26.6]
  Hospitalized, on non-invasive vent./high flow O2 | 4.4 [2.9 to 6.7] | 22.9 [12.1 to 39.0] | 7.4 [5.3 to 10.2] | 29.4 [16.8 to 46.2]
  Hospitalized, requiring supplemental oxygen | 24.1 [20.4 to 28.3] | 14.3 [6.3 to 29.4] | 21.0 [17.5 to 25.0] | 26.5 [14.6 to 43.1]
  Hospitalized, not on O2, requiring ongoing care | 11.9 [9.3 to 15.3] | 2.9 [0.5 to 14.5] | 9.8 [7.4 to 12.9] | 8.8 [3.0 to 23.0]
  Hospitalized, not requiring O2, no longer req care | 0.7 [0.2 to 1.9] | 0.0 [0.0 to 9.9] | 0.2 [0.0 to 1.3] | 0.0 [0.0 to 10.2]
  Not hospitalized, limit on activities/req home O2 | 56.0 [51.4 to 60.5] | 8.6 [3.0 to 22.4] | 57.8 [53.2 to 62.3] | 17.6 [8.3 to 33.5]
  Not hospitalized, no limitations on activities | 0.0 [0.0 to 0.8] | 0.0 [0.0 to 9.9] | 0.0 [0.0 to 0.9] | 0.0 [0.0 to 10.2]

37. Secondary Outcome: Percentage of Participants Reporting Each Severity Rating on an 8 Point Ordinal Scale at Day 11
Description: as for outcome 33
Time Frame: Day 11
Population: as for outcome 34
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 6
Number analyzed (Participants) | 452 | 35 | 448 | 34
percentage of participants
  Death at or before study visit | 0.9 [0.3 to 2.3] | 8.6 [3.0 to 22.4] | 1.6 [0.8 to 3.2] | 5.9 [1.6 to 19.1]
  Hospitalized, on invasive mech. vent. or ECMO | 3.1 [1.9 to 5.1] | 42.9 [28.0 to 59.1] | 2.7 [1.5 to 4.6] | 11.8 [4.7 to 26.6]
  Hospitalized, on non-invasive vent./high flow O2 | 2.9 [1.7 to 4.9] | 14.3 [6.3 to 29.4] | 2.9 [1.7 to 4.9] | 14.7 [6.4 to 30.1]
  Hospitalized, requiring supplemental oxygen | 10.0 [7.5 to 13.1] | 5.7 [1.6 to 18.6] | 12.7 [10.0 to 16.1] | 26.5 [14.6 to 43.1]
  Hospitalized, not on O2, requiring ongoing care | 5.8 [4.0 to 8.3] | 2.9 [0.5 to 14.5] | 5.8 [4.0 to 8.4] | 2.9 [0.5 to 14.9]
  Hospitalized, not requiring O2, no longer req care | 0.9 [0.3 to 2.3] | 2.9 [0.5 to 14.5] | 0.4 [0.1 to 1.6] | 0.0 [0.0 to 10.2]
  Not hospitalized, limit on activities/req home O2 | 73.9 [69.7 to 77.7] | 22.9 [12.1 to 39.0] | 70.5 [66.2 to 74.6] | 38.2 [23.9 to 55.0]
  Not hospitalized, no limitations on activities | 2.7 [1.5 to 4.6] | 0.0 [0.0 to 9.9] | 3.3 [2.0 to 5.5] | 0.0 [0.0 to 10.2]

38. Secondary Outcome: Percentage of Participants Reporting Each Severity Rating on an 8 Point Ordinal Scale at Day 15
Description: as for outcome 33
Time Frame: Day 15
Population: as for outcome 34
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 6
Number analyzed (Participants) | 452 | 35 | 448 | 34
percentage of participants
  Death at or before study visit | 1.3 [0.6 to 2.9] | 14.3 [6.3 to 29.4] | 2.0 [1.1 to 3.8] | 8.8 [3.0 to 23.0]
  Hospitalized, on invasive mech. vent. or ECMO | 2.2 [1.2 to 4.0] | 31.4 [18.6 to 48.0] | 3.1 [1.9 to 5.2] | 5.9 [1.6 to 19.1]
  Hospitalized, on non-invasive vent./high flow O2 | 1.1 [0.5 to 2.6] | 8.6 [3.0 to 22.4] | 1.8 [0.9 to 3.5] | 5.9 [1.6 to 19.1]
  Hospitalized, requiring supplemental oxygen | 6.0 [4.1 to 8.6] | 11.4 [4.5 to 26.0] | 6.0 [4.2 to 8.6] | 23.5 [12.4 to 40.0]
  Hospitalized, not on O2, requiring ongoing care | 3.1 [1.9 to 5.1] | 2.9 [0.5 to 14.5] | 2.5 [1.4 to 4.3] | 0.0 [0.0 to 10.2]
  Hospitalized, not requiring O2, no longer req care | 0.4 [0.1 to 1.6] | 0.0 [0.0 to 9.9] | 0.9 [0.3 to 2.3] | 0.0 [0.0 to 10.2]
  Not hospitalized, limit on activities/req home O2 | 53.1 [48.5 to 57.7] | 22.9 [12.1 to 39.0] | 52.5 [47.8 to 57.0] | 47.1 [31.5 to 63.3]
  Not hospitalized, no limitations on activities | 32.7 [28.6 to 37.2] | 8.6 [3.0 to 22.4] | 31.3 [27.1 to 35.7] | 8.8 [3.0 to 23.0]

39. Secondary Outcome: Percentage of Participants Reporting Each Severity Rating on an 8 Point Ordinal Scale at Day 22
Description: as for outcome 33
Time Frame: Day 22
Population: as for outcome 34
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 6
Number analyzed (Participants) | 452 | 35 | 448 | 34
percentage of participants
  Death at or before study visit | 2.2 [1.2 to 4.0] | 17.1 [8.1 to 32.7] | 2.5 [1.4 to 4.3] | 11.8 [4.7 to 26.6]
  Hospitalized, on invasive mech. vent. or ECMO | 1.8 [0.9 to 3.5] | 22.9 [12.1 to 39.0] | 1.6 [0.8 to 3.2] | 0.0 [0.0 to 10.2]
  Hospitalized, on non-invasive vent./high flow O2 | 0.7 [0.2 to 1.9] | 8.6 [3.0 to 22.4] | 0.2 [0.0 to 1.3] | 2.9 [0.5 to 14.9]
  Hospitalized, requiring supplemental oxygen | 4.0 [2.5 to 6.2] | 8.6 [3.0 to 22.4] | 4.2 [2.7 to 6.5] | 8.8 [3.0 to 23.0]
  Hospitalized, not on O2, requiring ongoing care | 1.8 [0.9 to 3.5] | 0.0 [0.0 to 9.9] | 1.6 [0.8 to 3.2] | 2.9 [0.5 to 14.9]
  Hospitalized, not requiring O2, no longer req care | 0.0 [0.0 to 0.8] | 0.0 [0.0 to 9.9] | 0.2 [0.0 to 1.3] | 0.0 [0.0 to 10.2]
  Not hospitalized, limit on activities/req home O2 | 48.0 [43.4 to 52.6] | 22.9 [12.1 to 39.0] | 49.6 [44.9 to 54.2] | 55.9 [39.5 to 71.1]
  Not hospitalized, no limitations on activities | 41.6 [37.1 to 46.2] | 20.0 [10.0 to 35.9] | 40.2 [35.7 to 44.8] | 17.6 [8.3 to 33.5]

40. Secondary Outcome: Percentage of Participants Reporting Each Severity Rating on an 8 Point Ordinal Scale at Day 29
Description: as for outcome 33
Time Frame: Day 29
Population: as for outcome 34
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 6
Number analyzed (Participants) | 452 | 35 | 448 | 34
percentage of participants
  Death at or before study visit | 3.1 [1.9 to 5.1] | 20.0 [10.0 to 35.9] | 2.9 [1.7 to 4.9] | 11.8 [4.7 to 26.6]
  Hospitalized, on invasive mech. vent. or ECMO | 1.8 [0.9 to 3.5] | 17.1 [8.1 to 32.7] | 1.6 [0.8 to 3.2] | 0.0 [0.0 to 10.2]
  Hospitalized, on non-invasive vent./high flow O2 | 0.7 [0.2 to 1.9] | 5.7 [1.6 to 18.6] | 0.0 [0.0 to 0.9] | 2.9 [0.5 to 14.9]
  Hospitalized, requiring supplemental oxygen | 2.7 [1.5 to 4.6] | 8.6 [3.0 to 22.4] | 2.0 [1.1 to 3.8] | 2.9 [0.5 to 14.9]
  Hospitalized, not on O2, requiring ongoing care | 1.3 [0.6 to 2.9] | 2.9 [0.5 to 14.5] | 0.7 [0.2 to 2.0] | 2.9 [0.5 to 14.9]
  Hospitalized, not requiring O2, no longer req care | 0.0 [0.0 to 0.8] | 0.0 [0.0 to 9.9] | 0.0 [0.0 to 0.9] | 0.0 [0.0 to 10.2]
  Not hospitalized, limit on activities/req home O2 | 65.9 [61.4 to 70.1] | 31.4 [18.6 to 48.0] | 67.2 [62.7 to 71.4] | 70.6 [53.8 to 83.2]
  Not hospitalized, no limitations on activities | 24.6 [20.8 to 28.7] | 14.3 [6.3 to 29.4] | 25.7 [21.8 to 29.9] | 8.8 [3.0 to 23.0]

41. Secondary Outcome: 14-day Participant Mortality
Description: The mortality rate was determined as the proportion of participants who died by study Day 15. The proportions reported are Kaplan-Meier estimates
Time Frame: Day 1 through Day 15
Population: The ITT population consists of all participants as randomized.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Remdesivir Plus Interferon Beta-1a | Remdesivir Plus Placebo
Number analyzed (Participants) | 487 | 482
Proportion of participants | 0.02 [0.01 to 0.03] | 0.02 [0.01 to 0.04]

42. Secondary Outcome: 28-day Participant Mortality
Description: The mortality rate was determined as the proportion of participants who died by study Day 29. The proportions reported are Kaplan-Meier estimates.
Time Frame: Day 1 through Day 29
Population: The ITT population consists of all participants as randomized
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Remdesivir Plus Interferon Beta-1a | Remdesivir Plus Placebo
Number analyzed (Participants) | 487 | 482
Proportion of participants | 0.05 [0.03 to 0.07] | 0.03 [0.02 to 0.06]

43. Secondary Outcome: Time to an Improvement of One Category Using an Ordinal Scale
Description: The ordinal scale is an assessment of the clinical status at the first assessment of a given study day. The scale is as follows: 8) Death; 7) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 6) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 5) Hospitalized, requiring supplemental oxygen; 4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 3) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 2) Not hospitalized, limitation on activities and/or requiring home oxygen; 1) Not hospitalized, no limitations on activities. Time to improvement by at least one category was determined for each participant.
Time Frame: Day 1 through Day 29
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 6
Number analyzed (Participants) | 452 | 35 | 448 | 34
Days | 12.0 [11.0 to 12.0] | 15.0 [7.0 to NA] — If no participants reach the upper limit of 95% CI of the KM estimator at the median then the upper limit of the median time to improvement of one category can not be estimated using the methodology described by Klein and Moeschberger (1997). | 12.0 [11.0 to 13.0] | 5.0 [4.0 to 7.0]
Statistical Analysis 1: Comparison: Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 vs Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5; Test type: Superiority; Cox Proportional Hazard = 1.04, 95% CI 2-sided [0.90 to 1.19]
Statistical Analysis 2: Comparison: Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 vs Remdesivir Plus Placebo in Baseline Ordinal Score 6; Test type: Superiority; Cox Proportional Hazard = 0.37, 95% CI 2-sided [0.21 to 0.66]

44. Secondary Outcome: Time to an Improvement of Two Categories Using an Ordinal Scale
Description: The ordinal scale is an assessment of the clinical status at the first assessment of a given study day. The scale is as follows: 1) Death; 2) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 3) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4) Hospitalized, requiring supplemental oxygen; 5) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 6) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 7) Not hospitalized, limitation on activities and/or requiring home oxygen; 8) Not hospitalized, no limitations on activities. Time to improvement by at least two categories was determined for each participant.
Time Frame: Day 1 through Day 29
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 6
Number analyzed (Participants) | 452 | 35 | 448 | 34
Days | 13.0 [NA to NA] — A large number of participants at the median estimate means there is little variability at the 50th percentile and the methodology described by Klein and Moeschberger (1997) is unable to compute a confidence interval. If no participants reach the upper limit of 95% CI of the KM estimator at 50%, the upper limit of the median time can not be estimated. | NA [14.0 to NA] — A large number of participants at the median estimate means there is little variability at the 50th percentile and the methodology described by Klein and Moeschberger (1997) is unable to compute a confidence interval. If no participants reach the upper limit of 95% CI of the KM estimator at 50%, the upper limit of the median time can not be estimated. Finally, if less than 50% of subjects improve by at least two categories then the median time cannot be estimated. | 13.0 [NA to NA] — A large number of participants at the median estimate means there is little variability at the 50th percentile and the methodology described by Klein and Moeschberger (1997) is unable to compute a confidence interval. If no participants reach the upper limit of 95% CI of the KM estimator at 50%, the upper limit of the median time can not be estimated. | 14.0 [13.0 to 19.0]
Statistical Analysis 1: Comparison: Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 vs Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5; Test type: Superiority; Cox Proportional Hazard = 1.04, 95% CI 2-sided [0.91 to 1.19]
Statistical Analysis 2: Comparison: Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 vs Remdesivir Plus Placebo in Baseline Ordinal Score 6; Test type: Superiority; Cox Proportional Hazard = 0.44, 95% CI 2-sided [0.24 to 0.82]

45. Secondary Outcome: Time to Discharge or to a National Early Warning Score (NEWS) of </= 2 and Maintained for 24 Hours, Whichever Occurs First
Description: The NEW score has demonstrated an ability to discriminate patients at risk of poor outcomes. This score is based on 7 clinical parameters (respiration rate, oxygen saturation, any supplemental oxygen, temperature, systolic blood pressure, heart rate, level of consciousness). The NEW Score is being used as an efficacy measure. The minimum score is 0, representing the better outcome, and the maximum value is 19, representing the worse outcome. The time to discharge or a NEWS of less than or equal to 2 was determined for each participant.
Time Frame: Day 1 through Day 29
Population: The modified intention-to-treat (mITT) population includes all participants who were randomized. mITT participants were classified by their randomized treatment assignment and their baseline ordinal score, which is not necessarily equivalent to the disease severity stratum to which the participant was randomized at enrollment, and restricted to those with a baseline NEWS score of 2 or greater.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 6
Number analyzed (Participants) | 356 | 33 | 354 | 34
Days | 4.0 [4.0 to 5.0] | NA [10.0 to NA] — If no participants reach the upper limit of 95% CI of the KM estimator at the median then the upper limit of the median time can not be estimated using the methodology described by Klein and Moeschberger (1997). Also, if less than 50% of participants discharge or reach a NEWS of </= 2 and maintain it for 24 Hours then the median time can not be estimated | 4.0 [4.0 to 5.0] | 9.0 [6.0 to 11.0]
Statistical Analysis 1: Comparison: Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 vs Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5; Test type: Superiority; Cox Proportional Hazard = 1.08, 95% CI 2-sided [0.93 to 1.26]
Statistical Analysis 2: Comparison: Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 vs Remdesivir Plus Placebo in Baseline Ordinal Score 6; Test type: Superiority; Cox Proportional Hazard = 0.39, 95% CI 2-sided [0.21 to 0.72]

46. Secondary Outcome: Time to Recovery for Patients With a Baseline Ordinal Score of 4 and 5
Description: Day of recovery is defined as the first day on which the subject satisfies one of the following three categories from the ordinal scale: 1) Not hospitalized, no limitations on activities; 2) Not hospitalized, limitation on activities and/or requiring home oxygen; 3) Hospitalized, not requiring supplemental oxygen and no longer requires ongoing medical care.
Time Frame: Day 1 through Day 29
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5
Number analyzed (Participants) | 452 | 448
Days | 5.0 [4.0 to 5.0] | 5.0 [4.0 to 5.0]
Statistical Analysis 1: Comparison: Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 vs Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5; Test type: Superiority; Cox Proportional Hazard = 1.04, 95% CI 2-sided [0.90 to 1.19]

47. Primary Outcome: Time to Recovery for Participants With Baseline Ordinal Score 4, 5 and 6 by Race
Description: as for outcome 1
Time Frame: Day 1 through Day 29
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Remdesivir Plus Interferon Beta-1a | Remdesivir Plus Placebo
Number analyzed (Participants) | 487 | 482
Days
  Asian: number analyzed (Participants) | 44 | 39
  Asian | 8.0 [6.0 to 9.0] | 8.0 [6.0 to 12.0]
  Black or African American: number analyzed (Participants) | 76 | 84
  Black or African American | 4.0 [4.0 to 5.0] | 4.0 [4.0 to 5.0]
  White: number analyzed (Participants) | 299 | 285
  White | 4.0 [4.0 to 5.0] | 5.0 [4.0 to 5.0]
  Other: number analyzed (Participants) | 68 | 74
  Other | 6.0 [5.0 to 7.0] | 5.0 [4.0 to 6.0]
Statistical Analysis 1: Comparison: Remdesivir Plus Interferon Beta-1a vs Remdesivir Plus Placebo; This analysis is for Asian participants; Test type: Superiority; Cox Proportional Hazard = 0.92, 95% CI 2-sided [0.59 to 1.45]
Statistical Analysis 2: Comparison: Remdesivir Plus Interferon Beta-1a vs Remdesivir Plus Placebo; This analysis is for Black and African American participants; Test type: Superiority; Cox Proportional Hazard = 0.92, 95% CI 2-sided [0.66 to 1.27]
Statistical Analysis 3: Comparison: Remdesivir Plus Interferon Beta-1a vs Remdesivir Plus Placebo; This analysis is for White participants; Test type: Superiority; Cox Proportional Hazard = 1.02, 95% CI 2-sided [0.86 to 1.21]
Statistical Analysis 4: Comparison: Remdesivir Plus Interferon Beta-1a vs Remdesivir Plus Placebo; This analysis is for Race of Other participants; Test type: Superiority; Cox Proportional Hazard = 0.84, 95% CI 2-sided [0.59 to 1.19]

48. Primary Outcome: Time to Recovery for Participants With Baseline Ordinal Score 4, 5 and 6 by Ethnicity
Description: as for outcome 1
Time Frame: Day 1 through Day 29
Population: The modified intention-to-treat (mITT) population includes all participants who were randomized and for whom Ethnicity was reported. mITT participants were classified by their randomized treatment assignment and their baseline ordinal score, which is not necessarily equivalent to the disease severity stratum to which the participant was randomized at enrollment.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Remdesivir Plus Interferon Beta-1a | Remdesivir Plus Placebo
Number analyzed (Participants) | 477 | 474
Days
  Not Hispanic or Latino: number analyzed (Participants) | 323 | 317
  Not Hispanic or Latino | 5.0 [4.0 to 5.0] | 5.0 [4.0 to 5.0]
  Hispanic or Latino: number analyzed (Participants) | 154 | 157
  Hispanic or Latino | 6.0 [5.0 to 7.0] | 5.0 [NA to NA] — A large number of participants at the median estimate means there is little variability at the 50th percentile and the methodology described by Klein and Moeschberger (1997) is unable to compute a confidence interval. Also, if less than 50% of participants recover then the median time can not be estimated.
Statistical Analysis 1: Comparison: Remdesivir Plus Interferon Beta-1a vs Remdesivir Plus Placebo; This analysis is for Not Hispanic or Latino participants; Test type: Superiority; Cox Proportional Hazard = 1.02, 95% CI 2-sided [0.86 to 1.19]
Statistical Analysis 2: Comparison: Remdesivir Plus Interferon Beta-1a vs Remdesivir Plus Placebo; This analysis is for Hispanic or Latino participants; Test type: Superiority; Cox Proportional Hazard = 0.83, 95% CI 2-sided [0.65 to 1.05]

49. Primary Outcome: Time to Recovery for Participants With Baseline Ordinal Score 4, 5 and 6 by Sex
Description: as for outcome 1
Time Frame: Day 1 through Day 29
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Remdesivir Plus Interferon Beta-1a | Remdesivir Plus Placebo
Number analyzed (Participants) | 487 | 482
Days
  Male: number analyzed (Participants) | 297 | 266
  Male | 5.0 [5.0 to 6.0] | 5.0 [5.0 to 6.0]
  Female: number analyzed (Participants) | 190 | 216
  Female | 4.5 [4.0 to 5.0] | 5.0 [4.0 to 5.0]
Statistical Analysis 1: Comparison: Remdesivir Plus Interferon Beta-1a vs Remdesivir Plus Placebo; This analysis is for Male participants; Test type: Superiority; Cox Proportional Hazard = 0.93, 95% CI 2-sided [0.78 to 1.10]
Statistical Analysis 2: Comparison: Remdesivir Plus Interferon Beta-1a vs Remdesivir Plus Placebo; This analysis is for Female participants; Test type: Superiority; Cox Proportional Hazard = 1.05, 95% CI 2-sided [0.86 to 1.29]

ADVERSE EVENTS:
Time Frame: Serious and Grade 3 and 4 non-serious adverse events were collected for 29 days after the first dose. Laboratory values were systematically assessed at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29. Treatment emergent and fatal AEs are reported.
Description: Given the severity of underlying illness, participants were expected to have many symptoms and abnormalities in vital signs and laboratory values. All Grade 3 and 4 AEs were captured as AEs in this trial. Grade 2 or higher, suspected drug-related hypersensitivity reaction or deep vein thrombosis of any grade was reported as an AE in this trial. All cause mortality was calculated for the ITT population, while SAEs and AEs reflect the as treated population.
Arm/Group | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 | Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5 | Remdesivir Plus Placebo in Baseline Ordinal Score 6
All-Cause Mortality (participants affected / at risk) | 14/452 | 7/35 | 13/448 | 4/34
Serious Adverse Events (participants affected / at risk) | 65/442 | 21/32 | 58/435 | 8/31
Other Adverse Events (participants affected / at risk) | 49/442 | 12/32 | 45/435 | 7/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 (N=442) | Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 (N=32) | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5 (N=435) | Remdesivir Plus Placebo in Baseline Ordinal Score 6 (N=31)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pulseless electrical activity (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 0 (0) | 1 (2) | 0 (0)
Septic shock (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Aspergillus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5) | 5 (5) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 5 (5) | 5 (5) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 19 (19) | 10 (10) | 21 (22) | 3 (3)
Diffuse alveolar damage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Distributive shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Embolism venous (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypertensive urgency (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Remdesivir Plus Interferon Beta-1a in Ordinal Score 4 and 5 (N=442) | Remdesivir Plus Interferon Beta-1a in Ordinal Score 6 (N=32) | Remdesivir Plus Placebo in Baseline Ordinal Score 4 and 5 (N=435) | Remdesivir Plus Placebo in Baseline Ordinal Score 6 (N=31)
Blood albumin decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 14 (16) | 4 (4) | 17 (18) | 1 (2)
Haemoglobin decreased (Investigations) | 5 (5) | 4 (6) | 7 (7) | 2 (2)
Lymphocyte count decreased (Investigations) | 30 (33) | 3 (4) | 27 (30) | 6 (6)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 1 (1) | 2 (2) | 4 (4)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2020-09-28): https://cdn.clinicaltrials.gov/large-docs/75/NCT04492475/Prot_001.pdf
  • Statistical Analysis Plan (2021-01-19): https://cdn.clinicaltrials.gov/large-docs/75/NCT04492475/SAP_002.pdf
  • Informed Consent Form (2020-11-13): https://cdn.clinicaltrials.gov/large-docs/75/NCT04492475/ICF_000.pdf